CLINICAL TRIAL: NCT04023474
Title: Role of Platelet-Rich Fibrin in the Healing of Regional and Free Flap Donor Sites for Head and Neck Surgery Patients: A Prospective Randomized Clinical Trial
Brief Title: Platelet-Rich Fibrin in the Healing of Regional and Free Flaps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201901618
Record Dates: First submitted 2019-07-12; First posted 2019-07-17 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Head and Neck Disorder; Free Flap
Keywords: Platelet-Rich Fibrin (PRF)
MeSH Terms: interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet Rich Fibrin (PRF) Group (Experimental): Patients randomized to this group will receive treatment with a PRF graft in clinic at the time any pertinent post-operative complication is identified.
  Interventions: Procedure: Platelet Rich Fibrin (PRF) Application
- No Platelet Rich Fibrin Group (No Intervention): Participants in the observational control group will be managed at the time of the complication by standard of care methods.

INTERVENTIONS:
Procedure: Platelet Rich Fibrin (PRF) Application — Platelet Rich Fibrin application to flap defect.
  Arms: Platelet Rich Fibrin (PRF) Group

SUMMARY:
Determine if the use of platelet-rich fibrin (PRF) versus historical treatment methods improves the post-operative management of healing complications from flap donor sites.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had surgery involving a microvascular free flap or a myocutaneous regional flap for head and neck reconstruction who develop one of the following donor site complications: wound dehiscence, wound margin breakdown or contraction resulting in healing by secondary intention, myocutaneous fistula formation, or incomplete coverage of the donor site by a skin graft placed in the operating room.

Exclusion Criteria:

* Patients under 18 years of age
* Patient's unable to participate in blood draw either due to medical compromise, inability to tolerate the procedure, or inability of the physician to successfully draw the blood at the time of appointment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Change in healing time at 3 months post-operative | Up to 3 months
  Improved healing of PRF patients compared to control group.

CONTACTS AND LOCATIONS:
Overall Officials: Salam Salman, MD, DDS, Principal Investigator — University of Florida
Locations (1):
- UF Health Jacksonville, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.